CLINICAL TRIAL: NCT02547961
Title: Chimeric Antigen Receptor-Modified T Cells for HER-2 Positive Recurrent and Metastatic Breast Cancer
Brief Title: Chimeric Antigen Receptor-Modified T Cells for Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Project terminated due to revision of local regulations
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Breast Cancer CAR-T 001
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; HER2; CAR-T cell
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HER2-CAR-T (Experimental): In interventional studies, participants are assigned to accept HER-2-targeting CAR T Cells infusion so that researchers can evaluate the effects and safety of the CAR-T cell.
  Interventions: Biological: HER-2-targeting CAR T Cells infusion
- No Intervention (No Intervention)

INTERVENTIONS:
Biological: HER-2-targeting CAR T Cells infusion — HER-2-targeting CAR t cells infusion in breast cancer
  Arms: HER2-CAR-T

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of HER2-CAR-T cell Infusion for advanced HER2 positive breast cancer.

DETAILED DESCRIPTION:
By enrolling patients with advanced HER2 positive breast cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of HER2-CAR-T cell infusion for advanced HER2 positive breast cancer.The CAR consists of a HER-2 targeting antibody scFv with two intracellular signaling domains derived from CD3 zeta and CD28. Autologous T cells will be gene-engineered with the CAR gene using a retrovirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Chemotherapy refractory Her2 positive breast cancer；
2. Relapsed patients after anti-Her2 using antibody or kinase inhibitor therapy；
3. Patients must be 18 years of age or older；
4. Patients must have an ECOG (Eastern Cooperative Oncology Group )performance status of 0-2；
5. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

Absolute neutrophil count greater than 1500/mm3. Platelet count greater than 100,000/mm3. Hemoglobin greater than 10g/dl (patients may receive transfusions to meet this parameter).

Total bilirubin < 1.5 times upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).

* Seronegative for HIV antibody.
* Seronegative for active hepatitis B, and seronegative for hepatitis C antibody.
* Patients must be willing to practice birth control during and for four months following treatment.NOTE:women of child-bearing age must have evidence of negative pregnancy test.
* Patients must be willing to sign an informed consent.

Exclusion Criteria:

* 1. Patients with uncontrolled hypertension (> 160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> New York Heart Association Class II), or myocardial infarction within 6 months of study will be excluded.

  2.Patients with any of the follo wing pulmonary function abnormalities will be excluded: FEV(forced expiratory volume), < 30% predicted; DLCO (diffusing capacity of lung for carbon monoxide) < 30% predicted (post-bronchodilator); Oxygen Saturation less than 90% on room air.

  3.Patients with severe liver and kidney dysfunction or consciousness disorders will be excluded.

  4.Pregnant and/or lactating women will be excluded. 5.Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.

  6.Patients with any type of primary immunodeficiencies will be excluded from the study.

  7.Patients requiring corticosteroids (other than inhaled) will be excluded. 8.Patients with history of T cell tumors will be excluded. 9.Patients who are participating or participated any other clinical trials in latest 30 days will be excluded.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events | 24weeks

SECONDARY OUTCOMES:
Tumor load | 24weeks
  Tumor load will be quantified with radiology, bone marrow and/or blood

OTHER OUTCOMES:
Progress free disease (PFS) | 1 year
Overall survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China